CLINICAL TRIAL: NCT01323647
Title: Immunogenicity and Safety of a Booster Dose of GlaxoSmithKline Biologicals' IPV (PoliorixTM) in Healthy Chinese Toddlers
Brief Title: Immunogenicity and Safety of Booster Dose of PoliorixTM Vaccine in Previously Vaccinated Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114306
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2017-05

CONDITIONS: Poliomyelitis
Keywords: IPV; PoliorixTM; China
MeSH Terms: conditions — Poliomyelitis | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (2):
- Group A (Experimental): Subjects in this group will receive the GSK Biologicals' IPV vaccine at 18 months of age. Subjects will also receive a dose of DTPa/Hib (Infanrix+Hib) as part of the local standard of care.
  Interventions: Biological: PoliorixTM; Biological: Infanrix+Hib
- Group B (Active Comparator): Subjects in this group will receive only a booster dose of GSK Biologicals' DTPa/Hib vaccine (Infanrix+Hib) as part of the local standard of care and will not be associated with any study endpoint.
  Interventions: Biological: Infanrix+Hib

INTERVENTIONS:
Biological: PoliorixTM — Single dose, intramuscular administration
  Arms: Group A
Biological: Infanrix+Hib — Single dose, intramuscular injection. Part of the local standard of care. No outcome measures associated.

SUMMARY:
This study aims to evaluate the persistence of anti-poliovirus antibodies in toddlers aged 18 months who were primed with oral polio vaccine (OPV) or inactivated polio vaccine (IPV) in the primary study. The study will also assess the immunogenicity and reactogenicity of a booster dose of IPV in subjects primed with three doses of IPV.

DETAILED DESCRIPTION:
All subjects will also receive a booster dose of GSK Biologicals' DTPa/Hib vaccine (Infanrix+Hib) at Day 0. This vaccine will be provided as part of the local standard of care and will not be associated with any study endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* Subjects who received the complete three-dose primary vaccination course in study NCT01021293.
* Healthy male or female toddlers 18 to 24 months of age at the time of Visit 1 (Day 0).
* Written informed consent obtained from the parent(s)/ Legally Acceptable Representative(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the booster dose of study vaccine(s), or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to Visit 1 (Day 0).
* Administration of immunoglobulins and/or any blood products within the 3 months preceding Visit 1 (Day 0) or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days of Visit 1 (Day 0) or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous booster vaccination against poliomyelitis or the disease since the conclusion visit of Study NCT01021293.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* Acute disease and/or fever at the time of enrolment.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 957 (Actual)
Dates: Start 2011-04-25; Primary Completion 2011-09-19 (Actual); Study Completion 2011-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- China (2):
  - GSK Investigational Site, Wuzhou, Guangxi
  - GSK Investigational Site, Mengshan Town

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Li R, Li CG, Li Y, Liu Y, Zhao H, Chen X, Kuriyakose S, Van Der Meeren O, Hardt K, Hezareh M, Roy-Ghanta S. Primary and booster vaccination with an inactivated poliovirus vaccine (IPV) is immunogenic and well-tolerated in infants and toddlers in China. Vaccine. 2016 Mar 14;34(12):1436-43. doi: 10.1016/j.vaccine.2016.02.010. Epub 2016 Feb 9. PMID 26873055
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114306 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114306 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114306 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114306 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114306 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114306 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Poliorix Group: Subjects previously primed with 3 doses of Poliorix™ vaccine in the primary study and who received a booster dose of Poliorix™ vaccine co-administered with Infanrix-Hib™ vaccine in the current study.
- Control Group: Subjects previously primed with 3 doses of Chinese oral poliovirus vaccine (OPV) in the primary study and who received a dose of Infanrix-Hib™ vaccine in the current study.
Period: Overall Study
Arm/Group | Poliorix Group | Control Group
Started | 470 | 487
Completed | 461 | 487
Not Completed | 9 | 0
Not completed — Migrated/moved from study area | 2 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Poliorix Group | Control Group | Total
Number analyzed (Participants) | 470 | 487 | 957
Age, Continuous [Mean (Standard Deviation); unit: Months] | 18.7 (0.93) | 18.8 (1.01) | 18.75 (0.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 227 | 461
  Male | 236 | 260 | 496
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Chinese heritage | 470 | 487 | 957

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroprotected for Poliovirus Types 1, 2 and 3 Antibodies Above the Cut-off Value
Description: A seroprotected subject was defined as a vaccinated subject whose antibody titer is greater than or equal to (≥) 8 Effective Dose 50 (ED50). This outcome measure concerns subjects in the Poliorix Group only.
Time Frame: One month after Poliorix™ booster vaccination.
Population: The According-to-Protocol (ATP) cohort for immunogenicity included all evaluable subjects who did not receive a product or present a medical condition leading to exclusion from an ATP analysis as listed in protocol and for whom data concerning immunogenicity outcome variables were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group
Number analyzed (Participants) | 456
Participants
  Anti-poliovirus 1 | 456
  Anti-poliovirus 2 | 456
  Anti-poliovirus 3 | 456

2. Primary Outcome: Number of Subjects Seroprotected for Poliovirus Types 1, 2 and 3 Antibodies Above the Cut-off Value
Description: A seroprotected subject was defined as a vaccinated subject whose antibody titer is greater than or equal to (≥) 8 ED50.
Time Frame: Before booster vaccination.
Population: The ATP cohort for antibody persistence included all subjects who completed the full 3-dose primary vaccination course in the primary study and have not received an additional dose of Poliorix vaccine since the primary study.Those who had no history of poliovirus infection,and for whom serological results were available at the persistence timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 470 | 484
Participants
  Anti-poliovirus 1 | 462 | 479
  Anti-poliovirus 2 | 445 | 482
  Anti-poliovirus 3 | 446 | 465

3. Primary Outcome: Antibody Titers Against Poliovirus Type 1, 2 and 3
Description: Antibody titers were summarized by geometric mean titers (GMTs) with their 95% confidence intervals (CIs). This outcome measure concerns subjects in the Poliorix Group only.
Time Frame: One month after Poliorix™ booster vaccination.
Population: The ATP cohort for immunogenicity included all evaluable subjects who did not receive a product or present a medical condition leading to exclusion from an ATP analysis as listed in protocol and for whom data concerning immunogenicity outcome variables were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Poliorix Group
Number analyzed (Participants) | 456
Titers
  Anti-poliovirus 1 | 3420.8 [3153.8 to 3710.5]
  Anti-poliovirus 2 | 1886.8 [1732.7 to 2054.5]
  Anti-poliovirus 3 | 5097 [4706.8 to 5519.6]

4. Primary Outcome: Antibody Titers Against Poliovirus Type 1, 2 and 3.
Description: Antibody titers were summarized by geometric mean titers (GMTs) with their 95% CIs.
Time Frame: Before booster vaccination.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 470 | 484
Titers
  Anti-poliovirus 1 | 97.6 [87.3 to 109.2] | 533.0 [468.0 to 607.0]
  Anti-poliovirus 2 | 87.8 [75.4 to 102.2] | 205.5 [185.6 to 227.5]
  Anti-poliovirus 3 | 109.7 [94.2 to 127.8] | 85.0 [76.1 to 95.0]

5. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = Cry when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site. This outcome measure concerns subjects in the Poliorix Group only.
Time Frame: Within 4-days (Days 0-3) post Poliorix™ booster vaccination.
Population: The Total Vaccinated cohort included all subjects, with booster dose administration documented, for whom data were available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group
Number analyzed (Participants) | 467
Participants
  Any Pain | 49
  Grade 3 Pain | 3
  Any Redness | 22
  Grade 3 Redness | 0
  Any Swelling | 11
  Grade 3 Swelling | 0

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed include drowsiness, irritability, loss of appetite and fever [defined as axillary temperature ≥ 37.1 degrees Celsius (°C)]. Any = occurence of any general symptom regardless of their intensity grade or relationship to study vaccine. Grade 3 drowsiness = drowsiness that prevented normal activities. Grade 3 fever = fever (axillary temperature) >39.0°C. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Related = symptom assessed by the investigator as causally related to the vaccination. This outcome measure concerns subjects in the Poliorix Group only.
Time Frame: Within 4-days (Days 0-3) post Poliorix™ booster vaccination.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group
Number analyzed (Participants) | 467
Participants
  Any Drowsiness | 59
  Grade 3 Drowsiness | 1
  Related Drowsiness | 59
  Any Irritability | 86
  Grade 3 Irritability | 2
  Related Irritability | 84
  Any Loss of appetite | 84
  Grade 3 Loss of appetite | 1
  Related Loss of appetite | 83
  Any temperature | 156
  Grade 3 temperature | 8
  Related temperature | 153

7. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an adverse event (AE) reported in addition to those solicited during the clinical study. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event. This outcome measure concerns subjects in the Poliorix Group only.
Time Frame: Within the 31-day (Days 0-30) follow-up period after the Poliorix™ booster vaccination.
Population: The Total Vaccinated cohort included all subjects, with booster dose administration documented and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group
Number analyzed (Participants) | 470
Participants | 22

8. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: During the entire study period (Day 0 to Month 1).
Population: The Total Cohort included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 470 | 487
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-Poliorix™ booster vaccination period; Unsolicited symptoms: during the 31-day (Days 0-30) post-Poliorix™ booster vaccination period. Serious Adverse Events (SAEs): during the entire study period (Day 0 to Month 1).
Description: Other (non-serious) adverse events were collected only for those subjects who had received a booster dose of Poliorix, i.e. Poliorix Group. No other (non-serious) adverse events data was collected for the Control Group.
Arm/Group | Poliorix Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/470 | 0/487
Serious Adverse Events (participants affected / at risk) | 0/470 | 1/487
Other Adverse Events (participants affected / at risk) | 202/470 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poliorix Group (N=470) | Control Group (N=487)
Pyrexia (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poliorix Group (N=470) | Control Group (N=0)
Decreased appetite (Metabolism and nutrition disorders) | 84 (84) | 0 (0)
Irritability (Psychiatric disorders) | 86 (86) | 0 (0)
Pain (General disorders) | 49 (49) | 0 (0)
Pyrexia (General disorders) | 157 (158) | 0 (0)
Somnolence (Nervous system disorders) | 59 (59) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.